CLINICAL TRIAL: NCT02993770
Title: Comparison of Endonasal-Endoscopic Dacryocystorhinostomy Versus External Dacryocystorhinostomy
Brief Title: Endo-nasal Endoscopic DCR and External-DCR in Primary Nasolacrimal Duct Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR.TUMS.REC.1394.853
Record Dates: First submitted 2016-09-10; First posted 2016-12-15 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2019-09

CONDITIONS: Primary Acquired Nasolacrimal

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Endoscopic DCR (Experimental): Endoscopic DCR will be performed by a single ophthalmic plastic surgeon expert in endoscopic surgery (F.P.) with a modified powered endonasal endoscopic technique described by Wormold.
  Interventions: Procedure: Endoscopic DCR; Procedure: External DCR
- External DCR (Active Comparator): External DCR will be performed in a conventional mannervia a nasal side straight skin incision 1 cm medial to medial canthal area, 1 cm long, then orbicularis oculi muscle will be separated using blunt dissection to expose the periosteum overlying and medial to the anterior lacrimal crest
  Interventions: Procedure: Endoscopic DCR; Procedure: External DCR

INTERVENTIONS:
Procedure: Endoscopic DCR — Endonasal endoscopic technique as described by Wormold et al.
Procedure: External DCR — External DCR

SUMMARY:
All patients with epiphora or eye discharge that admitted to our ophthalmic plastic clinic in Farabi hospital will be systemically evaluated. Those with confirmed diagnosis of primary nasolacrimal duct obstruction (PANDO) that need DCR by one senior ophthalmic plastic consultant, will be randomly assigned to one of the 2 treatment groups: Group 1 External DCR and group 2 En-DCR. Diagnosis of PANDO will be based on the presence of positive regurgitation test or irrigation test or dacryocystography (DCG) . All patients will undergo comprehensive ophthalmology examinations including best corrected visual acuity (BCVA), relative afferent pupillary defect (RAPD), slit lamp anterior segment evaluation, dilated fundoscopy with 78 D lens. Past history and review os systems will be elicited for medications, past or intercurrent dacryocystitis,trauma,past ocular and sinus surgeries, epiphora, discharge, ocular diseases, sinus/nasal diseases, diabetes mellitus, organ transplant, immunosuppressive drugs and immunodeficiency disorders.

All operations will be performed under general or local anesthesia, based on patient and surgeon preferences.

Surgical Technique:

All En-DCR surgeries will be performed by a single ophthalmic plastic surgeon expert in endoscopic surgery (F.P.) with a modified powered endonasal endoscopic technique described by Wormold.

Using a 0 degree 4-mm endonasal endoscope nasal mucoperiosteum in the area of the lacrimal sac will be incised and elevated. Then rhinostomy will be made using forceps, exposing lacrimal sac. Lacrimal sac will be opened and a Crawford silicone tube will be passed through puncta into nasal cavity and stabilized and will be kept for 2 months. After operation patients will receive nasal beclomethasone twice daily for 2 weeks, nasal drop phenylephrine 0.25% four times daily and ophthalmic drop fluorometholone and Levofloxacin four times daily for one week.

External DCR will be performed in a conventional manner [2]via a nasal side straight skin incision 1 cm medial to medial canthal area, 1 cm long, then orbicularis oculi muscle will be separated using blunt dissection to expose the periosteum overlying and medial to the anterior lacrimal crest. After incision of the periosteum, an osteotomy approximately 10 mm in diameter will be prepared. The lacrimal sac and then nasal mucosa will be opened by an "H" incision to form maximal anterior flaps. A Bodkin tube will be passed through puncta into nasal cavity of stabilized by multiple square knots at the end. The small posterior flaps will be cut and excised and anterior flaps will be sutured together with 2 or 3 6-0 vicryl sutures. The periosteum, orbicularis oculi muscle, will be sutured by 6-0 vicryl sutures. Skin will be sutured by Nylon 6-0 by interrupted style in the standard manner. Nasal packing will not be placed. All Ext-DCR operations will be performed by one of the two expert ophthalmic plastic surgeons (F.P and A.K.).

The amount of bleeding will be estimated and recorded by the subtracting the total suction reservoir from the amount of irrigated fluid through syringe during operation. Time of operation will be estimated and recorded from the time of anesthetics injection to removing the drape.

One week after operation patients will be asked to report post-operative pain and discomfort by visual analogue score scale (0-10).

27 Seven days after operation skin sutures of patients in group 2 will be removed if skin is healed, and complications, if any, will be detected and recorded in the special data sheets. Nasal bleeding, medial canthal swelling and erythema, ocular surface fluorescein staining and any complications will be detected and recorded. Dye disappearance test (DDT) will be checked and recorded. Epiphora will be recorded according to modified Munk epiphora staging scale.

Two months after operation, ocular surface will be checked by fluorescein for staining of cornea and conjunctiva. Then silicone tube will be removed. epiphora will be recorded according to our staging system. Dye disappearance test (DDT) and Fluorescein Dynamic Dye test (FDDT) and irrigation test, epiphora and skin scar by visual analogue scale (VAS) visual analogue scale will be checked in months 2, 6, 12, 18 and after operation. Satisfaction will be checked 2 mo and 18 mo after operation by VAS. Any grade of daily epiphora or return of fluid>20% through opposite punctum in irrigation test or negative FDDT (absence of fluid passage) will be regarded as functional or anatomic failure, respectively. Any complication will be recorded in the specific forms.

All pre-operative and post-op examinations will be performed by a masked senior ophthalmology resident subjective data will be checked and recorded by a trained nurse

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 year.
2. Diagnosis of PANDO (primary acquired nasolacrimal duct obstruction) if each one of the following exist:

1) Regurgitation of pus/mucous by pressure on lacrimal sac. 2) Return of pus/mucous fluid by irrigation test through one lacrimal punctum. 3) Dacryocystography or lacrimal scintigraphy compatible with nasolacrimal duct obstruction.

3. Absence of secondary causes of nasolacrimal duct obstruction (NLDO) such as nasal and sinuses diseases, inflammatory and neoplastic lesions involving the lacrimal drainage system, nasolacrimal trauma.

Exclusion Criteria:

1. Punctal/Canalicular obstruction.
2. Use of anti-coaggulation medications [aspirin, NSAIDS (non-steroidal anti-inflammatory drugs), Warfarin] within 3-10 days before surgery.
3. Handicap/mental retardation.
4. Pregnant women.
5. Patients with Immunodeficient status (AIDS, use of immunosuppressive medications, leukemia, lymphoma,..).
6. Nasal inflammatory disease (rhinitis, allergies).
7. Granulomatous diseases such as Wegeners, Sarcoidosis, etc.
8. History of past lacrimal surgery.
9. Traumatic NLDO.
10. Follow up less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Anatomic success rate of endonasal endoscopic- DCR (En-DCR) with traditional external-DCR (Ext-DCR) in patients with PANDO | 12 months after operation.
  anatomic patency of lacrimal drainage
Functional success rate endonasal endoscopic- DCR (En-DCR) with traditional external-DCR (Ext-DCR) in patients with PANDO | 12 months after operation.
  absence of epiphora and discharge
general success rate | 12 months after operation.
  anatomic patency of lacrimal drainage+ Functional such (absence of epiphora and discharge )

SECONDARY OUTCOMES:
Complications of operation | 12 months after operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Farabi Hospital, Tehran University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided